CLINICAL TRIAL: NCT04580589
Title: Investigation of Genetic Variations on Patients With Adverse Events While on Direct Oral Anticoagulants (DOACs)
Brief Title: DOAC ADRs Retrospective Study on Genetic Variations
Acronym: DARES1
Status: Completed | Type: Observational
Sponsor: Cipherome, Inc. (Industry)
Collaborators: Santa Clara Valley Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: C02-001 SC003
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Drug-Related Side Effects and Adverse Reactions; Treatment Failure
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood DNA sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adverse Drug Reaction on DOAC: Participants on Direct Oral Anti-coagulants (DOACs) who experience major bleeding or clinically relevant non-major bleeding per International Society of Thrombosis and Haemostasis criteria. This is an observational study, so there will be no intervention.
- Treatment Failure on DOAC: Participants on Direct Oral Anti-coagulants (DOACs) who experience treatment failure (e.g., recurrent MI, systemic embolism, ischemic stroke, etc.). This is an observational study, so there will be no intervention.
- Case Control: Participants on Direct Oral Anti-coagulants (DOACs) who experience neither major bleeding or treatment failure.

SUMMARY:
The purpose of this study is to see if the participant's genetic profile and clinical factors (age, drug dose, etc.) affect drug outcomes (i.e. serious bleeding) that the participant may have experienced since taking the drug (direct oral anticoagulant) for preventing blood clots from forming in the blood vessels.

DETAILED DESCRIPTION:
Genes can have variants or mutations that can increase the participant's risk for bleeding when receiving a direct oral anticoagulant (DOACs). The investigators will be studying participants on DOACs who have had bleeding and also participants who are on DOACs who did not have bleeding (control group). The goal of the study is to determine the accuracy of Cipherome's Drug Safety Score (DSS) in it's ability to predict adverse drug reactions (ADRs). A DSS score ranges from 0 to 1, with scores less than 0.3 correlated with a higher risk of ADRs and scores more than 0.7 correlated with a lower risk of ADRs. The participant's DSS score will be compared with the actual clinical outcome using a statistical test to determine the accuracy of the DSS.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient 18 years and older, who experienced major bleeding, clinically relevant non major bleeding or treatment failure while taking a DOAC during the study time frame and is able to provide informed consent. Control patients will be recruited from all adult patients who are on DOAC therapy.

Exclusion Criteria:

* Failure to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any adult patient 18 years and older, who experienced major bleeding, clinically relevant non major bleeding or treatment failure while taking a DOAC during the study time frame and is able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Major bleeding event during DOAC therapy | Within 1 year of DOAC therapy initiation
  * Reduction in hemoglobin of at least 2 g/dL
  * Blood loss requiring transfusion of at least 2 units of whole blood or erythrocytes
  * Critical anatomical sites of bleeding: intramuscular with compartment syndrome, intracranial, intraspinal, retroperitoneal, intraocular, pericardial, and atraumatic intra-articular bleeding.
  * Bleeding leading to death
Clinically relevant non-major bleeding | Within 1 year of DOAC therapy initiation
  * Hospital admission for bleeding, or
  * Physician guided medical or surgical treatment for bleeding, or
  * Change in antithrombotic therapy (including interruption or discontinuation of study drug).

SECONDARY OUTCOMES:
Thromboembolic events | Within 1 year of DOAC therapy initiation
  Thromboembolic events including, but not limited to: deep vein thrombosis, pulmonary embolism, ischemic stroke, transient ischemic attack, arterial thrombosis, or other thromboembolic event

OTHER OUTCOMES:
Discovery of novel genetic variants | Within 1 year of DOAC therapy initiation
  To discover novel pharmacogenomic variants associated with DOAC metabolism. The investigators will be conducting whole genome sequencing to determine novel variants found in individuals with major bleeding or treatment failures.

CONTACTS AND LOCATIONS:
Overall Officials: Dayani Nualles-Percy, MD, Principal Investigator — Santa Clara Valley Medical Center; Clifford Wang, MD, Study Director — Santa Clara Valley Medical Center
Locations (1):
- Santa Clara Valley Medical Center, Santa Clara, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Wysowski DK, Nourjah P, Swartz L. Bleeding complications with warfarin use: a prevalent adverse effect resulting in regulatory action. Arch Intern Med. 2007 Jul 9;167(13):1414-9. doi: 10.1001/archinte.167.13.1414. PMID 17620536
- [Background] Zareh M, Davis A, Henderson S. Reversal of warfarin-induced hemorrhage in the emergency department. West J Emerg Med. 2011 Nov;12(4):386-92. doi: 10.5811/westjem.2011.3.2051. PMID 22224125
- [Background] Kirley K, Qato DM, Kornfield R, Stafford RS, Alexander GC. National trends in oral anticoagulant use in the United States, 2007 to 2011. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):615-21. doi: 10.1161/CIRCOUTCOMES.112.967299. Epub 2012 Sep 4. PMID 22949490
- [Background] Bauer KA. Pros and cons of new oral anticoagulants. Hematology Am Soc Hematol Educ Program. 2013;2013:464-70. doi: 10.1182/asheducation-2013.1.464. PMID 24319220
- [Background] Kanuri SH, Kreutz RP. Pharmacogenomics of Novel Direct Oral Anticoagulants: Newly Identified Genes and Genetic Variants. J Pers Med. 2019 Jan 17;9(1):7. doi: 10.3390/jpm9010007. PMID 30658513
- [Background] Sennesael AL, Larock AS, Douxfils J, Elens L, Stillemans G, Wiesen M, Taubert M, Dogne JM, Spinewine A, Mullier F. Rivaroxaban plasma levels in patients admitted for bleeding events: insights from a prospective study. Thromb J. 2018 Nov 12;16:28. doi: 10.1186/s12959-018-0183-3. eCollection 2018. PMID 30455596
- [Background] Ing Lorenzini K, Daali Y, Fontana P, Desmeules J, Samer C. Rivaroxaban-Induced Hemorrhage Associated with ABCB1 Genetic Defect. Front Pharmacol. 2016 Dec 19;7:494. doi: 10.3389/fphar.2016.00494. eCollection 2016. PMID 28066243
- [Background] Ueshima S, Hira D, Kimura Y, Fujii R, Tomitsuka C, Yamane T, Tabuchi Y, Ozawa T, Itoh H, Ohno S, Horie M, Terada T, Katsura T. Population pharmacokinetics and pharmacogenomics of apixaban in Japanese adult patients with atrial fibrillation. Br J Clin Pharmacol. 2018 Jun;84(6):1301-1312. doi: 10.1111/bcp.13561. Epub 2018 Apr 16. PMID 29457840
- [Background] Shi J, Wang X, Nguyen JH, Bleske BE, Liang Y, Liu L, Zhu HJ. Dabigatran etexilate activation is affected by the CES1 genetic polymorphism G143E (rs71647871) and gender. Biochem Pharmacol. 2016 Nov 1;119:76-84. doi: 10.1016/j.bcp.2016.09.003. Epub 2016 Sep 8. PMID 27614009
- [Background] Dimatteo C, D'Andrea G, Vecchione G, Paoletti O, Cappucci F, Tiscia GL, Buono M, Grandone E, Testa S, Margaglione M. Pharmacogenetics of dabigatran etexilate interindividual variability. Thromb Res. 2016 Aug;144:1-5. doi: 10.1016/j.thromres.2016.05.025. Epub 2016 May 26. PMID 27261537
- [Background] Sychev DA, Levanov AN, Shelekhova TV, Bochkov PO, Denisenko NP, Ryzhikova KA, Mirzaev KB, Grishina EA, Gavrilov MA, Ramenskaya GV, Kozlov AV, Bogoslovsky T. The impact of ABCB1 (rs1045642 and rs4148738) and CES1 (rs2244613) gene polymorphisms on dabigatran equilibrium peak concentration in patients after total knee arthroplasty. Pharmgenomics Pers Med. 2018 Jul 25;11:127-137. doi: 10.2147/PGPM.S169277. eCollection 2018. PMID 30100750
- [Background] 1000 Genomes Project Consortium; Auton A, Brooks LD, Durbin RM, Garrison EP, Kang HM, Korbel JO, Marchini JL, McCarthy S, McVean GA, Abecasis GR. A global reference for human genetic variation. Nature. 2015 Oct 1;526(7571):68-74. doi: 10.1038/nature15393. PMID 26432245
- [Background] Beckman MG, Hooper WC, Critchley SE, Ortel TL. Venous thromboembolism: a public health concern. Am J Prev Med. 2010 Apr;38(4 Suppl):S495-501. doi: 10.1016/j.amepre.2009.12.017. PMID 20331949
- [Background] Schulman S, Kearon C, Kakkar AK, Schellong S, Eriksson H, Baanstra D, Kvamme AM, Friedman J, Mismetti P, Goldhaber SZ; RE-MEDY Trial Investigators; RE-SONATE Trial Investigators. Extended use of dabigatran, warfarin, or placebo in venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):709-18. doi: 10.1056/NEJMoa1113697. PMID 23425163